CLINICAL TRIAL: NCT03693313
Title: The Effect of CrossFit Kids on Social Skills in Children With Autism Spectrum Disorder (CrossFit KAMP)
Acronym: CrossFit KAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1235533
Record Dates: First submitted 2018-06-06; First posted 2018-10-02 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD, Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Wait List Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CrossFit KAMP Group 1 (Experimental): 14 weeks of CrossFit Kids exercise program
  Interventions: Behavioral: CrossFit Kids exercise program
- CrossFit KAMP Wait-list Group (Active Comparator): Waitlist group that waits 14 weeks while group 1 does exercise program. After first 14 weeks will then participate in 14 weeks of CrossFit Kids exercise program
  Interventions: Behavioral: CrossFit Kids exercise program

INTERVENTIONS:
Behavioral: CrossFit Kids exercise program — Participants will be actively participating in a 14 week twice weekly CrossFit Kids exercise program.

SUMMARY:
The Centers for Disease Control and Prevention estimates that 1 in 59 U.S. children have been diagnosed with an autism spectrum disorder (ASD). Peer relationships, social skills, and repetitive behaviors are a challenge for those with ASD. Exercise in the ASD population has been examined as a means to improve some of these challenges for children with ASD. This research study will try to see if a structured exercise program called CrossFit Kids can help with these challenges. This study is potentially beneficial in developing an exercise program for children with ASD that can help promote social skill development, reduce stereotypical behaviors, and provide overall health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Autism Spectrum Disorder
* Full Scale IQ >80 on standardized testing
* English speaking
* Parents must be able to bring children to class twice a week for 14 weeks.

Exclusion Criteria:

* Non-English speaking
* Medical condition or physical impairment precluding them from safely participating in classes (eg. spastic quadriplegic cerebral palsy, critical congenital heart disease, uncontrolled asthma, uncontrolled seizure disorder, etc.)

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Improvement in social skills in children with ASD | 40 weeks
  The Social Responsiveness Scale, 2nd edition is a parent questionnaire that describes difficulties in socialization, communication, and repetitive/restricted interests. The SRS includes parent and teacher evaluations and provides quantitative subscales that can distinguish the presence of ASD from other child psychiatric conditions. Scale will be administered pre CrossFit Kids intervention, after the 14 weeks of CrossFit Kids and then 8 weeks after the intervention of CrossFit Kids. Total T-score ranges 59 and below=within normal limits; 60-65 =mild range, 66-75 =moderate range, 76 or higher = severe range. Lower T-score means participant is less affected.
Improvement in behavioral symptoms in children with ASD | 40 weeks
  The Behavioral Symptoms Index on the Behavioral Assessment System for Children, 3rd edition (BASC-3). Parent report is a parent rating scale that will be used as a general behavioral screen for comorbidities (hyperactivity, other externalizing behaviors, depression, etc.). Scale will be administered pre CrossFit Kids intervention, after the 14 weeks of CrossFit Kids and then 8 weeks after the intervention of CrossFit Kids. T scores are as follows 60 or less= within normal limits, 60-70 =at risk, 70 or higher= clinically significant. Lower T-score means less behavioral symptoms.
Improvement in repetitive behaviors in children with ASD | 40 weeks
  The Repetitive Behavior Scale Revised (RBS-R) is a parent questionnaire that measures six subscales of repetitive behavior including: Stereotyped Behavior, Self-injurious Behavior, Compulsive Behavior, Routine Behavior, Sameness Behavior, and Restricted Behavior in those with ASD. Scale will be administered pre CrossFit Kids intervention, after the 14 weeks of CrossFit Kids and then 8 weeks after the intervention of CrossFit Kids. Higher total scores on repetitive behavior scale are associated with higher amounts of repetitive behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States